CLINICAL TRIAL: NCT04909853
Title: A PHASE 1, NON-RANDOMIZED, OPEN-LABEL STUDY TO ASSESS THE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF PF-07321332 BOOSTED WITH RITONAVIR IN ADULT PARTICIPANTS WITH RENAL IMPAIRMENT AND IN HEALTHY PARTICIPANTS WITH NORMAL RENAL FUNCTION.
Brief Title: Renal Impairment Study of PF-07321332 Boosted With Ritonavir in Adult Participants With Renal Impairment and in Healthy Participants With Normal Renal Function.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C4671011
Record Dates: First submitted 2021-05-29; First posted 2021-06-02 (Actual); Results first posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2022-09

CONDITIONS: Renal Impairment
Keywords: SARS-CoV-2; COVID-19
MeSH Terms: conditions — Renal Insufficiency; COVID-19 | interventions — nirmatrelvir and ritonavir drug combination; nirmatrelvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-07321332 (Experimental): PF 07321332/ritonavir
  Interventions: Drug: PF-07321332/ritonavir

INTERVENTIONS:
Drug: PF-07321332/ritonavir — PF-07321332 in combination with the PK boosting agent, ritonavir, being developed for the treatment of COVID-19
  Other Names: PF-07321332

SUMMARY:
This is a Phase 1, non-randomized, open-label, 2-part study to investigate the effect of renal impairment on the pharmacokinetics (PK), safety and tolerability of a single oral dose of PF-07321332 in combination with the PK boosting agent ritonavir. Participants will be selected and categorized into normal renal function or renal impairment groups based on their estimated glomerular filtration rate. Part 1: will be conducted in approximately 24 participants (approximately 8 per group) with stable mild or moderate renal impairment and a control group of participants with normal renal function. Part 2 will be conducted in approximately 8 participants with stable severe renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, non-smoker and/or light smoker
* Have a diagnosis of stable renal impairment
* Meet the following estimated glomerular filtration rate (eGFR) criteria during the screening period (based on 2 Screening visits) based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation:

  * Mild renal impairment: eGFR between 60 - 89 mL/min.
  * Moderate renal impairment: eGFR ≥30 mL/min and <60 mL/min.
  * Severe renal impairment: eGFR <30 mL/min, but not requiring hemodialysis.
  * Normal renal function: eGFR ≥90 mL/min

Renal impairment participants:

* Any form of renal impairment except acute nephritic syndrome (participants with history of previous nephritic syndrome but in remission can be included).
* Good general health commensurate with the population with chronic kidney disease (renal impairment).
* Stable concomitant drug regimen for the management of individual participant's medical conditions, so long as they are considered necessary for the welfare of the study participants (eg, standard therapy for underlying diseases), and are not contraindicated with study drug, and are unlikely to interfere with the PK of study drug.

Healthy participants with normal renal function:

* No clinically relevant abnormalities identified by a detailed medical history, full physical examination, including temperature, blood pressure (BP) and pulse rate measurement, 12 lead ECG and clinical laboratory tests.
* Demographically comparable to the group of participants with impaired renal function.

  * Each participant's body weight within ±15 kg of the mean body weight of renal impairment group.
  * Each participant's age within ±10 years of the mean age of the renal impairment group.

Exclusion Criteria:

* Positive test result for SARS-CoV-2 infection at the time of screening or Day -1.
* History of HIV infection, hepatitis B, or hepatitis C; positive testing at screening for HIV, HBsAg, HBcAb, or HCVAb. As an exception a positive HBsAb test due to Hepatitis B vaccination is allowed.
* Renal transplant recipients.
* Urinary incontinence without catheterization
* Any condition possibly affecting drug absorption (eg, prior bariatric surgery, gastrectomy, cholecystectomy, appendectomy).
* Participants who have been vaccinated with COVID-19 vaccines within the past 2 weeks of dosing, or are to be vaccinated with these vaccines at any time during the study.
* A positive urine drug test, for illicit drugs, at Screening
* aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level >2 × upper limit of normal (ULN)
* Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is≤ ULN.
* History of sensitivity reactions to ritonavir or any of the formulation components of PF 07321332 or ritonavir.
* Female participants of childbearing potential who are unwilling or unable to use highly effective methods of contraception as outlined in Section 5.3.4 for the duration of the study and for at least 28 days after the administration of investigational product, pregnant female participants, female participants planning to become pregnant during the duration of the study until 28 days after the administration of investigational product, breastfeeding female participants.

Renal impairment participants:

* Participants requiring hemodialysis and/or peritoneal dialysis
* Participants with other clinically significant disease that may affect the safety of the participant or that may affect the PK of PF-07321332. Participants with any significant hepatic, cardiac, or pulmonary disease or participants who are clinically nephrotic.

Healthy participants with normal renal function:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Screening supine BP >140 mm Hg (systolic) or >90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is >140 mm Hg (systolic) or >90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Orange County Research Center, Tustin, California
  - Investigational Drug Services (IDS) University of Miami Hospitals and Clinics, Miami, Florida
  - University of Miami Division of Clinical Pharmacology, Miami, Florida
  - Genesis Clinical Research, LLC, Tampa, Florida
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Toussi SS, Neutel JM, Navarro J, Preston RA, Shi H, Kavetska O, LaBadie RR, Binks M, Chan PLS, Demers N, Corrigan B, Damle B. Pharmacokinetics of Oral Nirmatrelvir/Ritonavir, a Protease Inhibitor for Treatment of COVID-19, in Subjects With Renal Impairment. Clin Pharmacol Ther. 2022 Oct;112(4):892-900. doi: 10.1002/cpt.2688. Epub 2022 Jul 5. PMID 35712797
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study had 2 parts, Part 1 and 2. Enrollment were separate for both the parts. A total of 35 participants (27 in Part 1 and 8 in Part 2) were enrolled in the study of which 34 participants received the study treatment.
Pre-assignment Details: Participants were grouped on the basis of severity of renal impairment. Severity was evaluated using estimated glomerular filtration rate (eGFR) in milliliter per minute (mL/min) based on chronic kidney disease-epidemiology collaboration (CKD-EPI) formula. Following were the classifications, a) Normal: eGFR greater than or equal to (>=) 90 mL/min, b) Mild: eGFR 60 to less than (<) 90 mL/min, c) Moderate: eGFR >= 30 to <60 mL/min and d) Severe: eGFR <30 mL/min and not requiring dialysis.
Groups:
- Part 1: Normal Renal Function: Participants with normal renal function received PF-07321332 100 milligram (mg) single oral dose on Day 1 of Part 1 of the study. Participants were administered with pharmacokinetic boosting agent ritonavir 100 mg orally on Day -1 at -12 hours, Day 1 at 0 hours and 12 hours, and Day 2 at 24 hours, relative to PF-07321332 dosing in Part 1 of the study. Participants were followed-up to maximum of 35 days after the last administration of ritonavir or from the time of early termination/discontinuation.
- Part 1: Mild Renal Impairment: Participants with mild renal function received PF-07321332 100 mg single oral dose on Day 1 of Part 1 of the study. Participants were administered with pharmacokinetic boosting agent ritonavir 100 mg orally on Day -1 at -12 hours, Day 1 at 0 hours and 12 hours, and Day 2 at 24 hours, relative to PF-07321332 dosing in Part 1 of the study. Participants were followed-up to maximum of 35 days after the last administration of ritonavir or from the time of early termination/discontinuation.
- Part 1: Moderate Renal Impairment: Participants with moderate renal function received PF-07321332 100 mg single oral dose on Day 1 of Part 1 of the study. Participants were administered with pharmacokinetic boosting agent ritonavir 100 mg orally on Day -1 at -12 hours, Day 1 at 0 hours and 12 hours, and Day 2 at 24 hours, relative to PF-07321332 dosing in Part 1 of the study. Participants were followed-up to maximum of 35 days after the last administration of ritonavir or from the time of early termination/discontinuation.
- Part 2: Severe Renal Impairment: Participants with severe renal function received PF-07321332 100 mg single oral dose on Day 1 of Part 2 of the study. Participants were administered with pharmacokinetic boosting agent ritonavir 100 mg orally on Day -1 at -12 hours, Day 1 at 0 hours and 12 hours, and Day 2 at 24 hours, relative to PF-07321332 dosing in Part 2 of the study. Participants were followed-up to maximum of 35 days after the last administration of ritonavir or from the time of early termination/discontinuation.
Period: Part 1
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Started | 10 | 8 | 9 | 0
Treated | 10 | 8 | 8 | 0
Completed | 10 | 8 | 8 | 0
Not Completed | 0 | 0 | 1 | 0
Not completed — Assigned but not treated | 0 | 0 | 1 | 0
Period: Part 2
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Started | 0 (Participants from Part 1 did not enter in Part 2. Enrollment was separate for Part 1 and 2.) | 0 (Participants from Part 1 did not enter in Part 2. Enrollment was separate for Part 1 and 2.) | 0 (Participants from Part 1 did not enter in Part 2. Enrollment was separate for Part 1 and 2.) | 8 (Enrollment was separate for Part 1 and 2.)
Completed | 0 | 0 | 0 | 7
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Groups:
- Part 1: Normal Renal Function: Participants with normal renal function received PF-07321332 100 mg single oral dose on Day 1 of Part 1 of the study. Participants were administered with pharmacokinetic boosting agent ritonavir 100 mg orally on Day -1 at -12 hours, Day 1 at 0 hours and 12 hours, and Day 2 at 24 hours, relative to PF-07321332 dosing in Part 1 of the study. Participants were followed-up to maximum of 35 days after the last administration of ritonavir or from the time of early termination/discontinuation.
- Total: Total of all reporting groups
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment | Total
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.1 (3.03) | 63.8 (9.07) | 62.0 (8.57) | 62.1 (9.46) | 62.2 (7.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 2 | 11
  Male | 7 | 5 | 5 | 6 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 0 | 4 | 9
  Not Hispanic or Latino | 6 | 7 | 8 | 4 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 6 | 2 | 12
  White | 7 | 6 | 2 | 6 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-07321332
Time Frame: Part 1 and Part 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose on Day 1
Population: The pharmacokinetic (PK) parameter analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Number analyzed (Participants) | 10 | 8 | 8 | 8
Nanogram per milliliter | 1600 (31) | 2077 (29) | 2210 (17) | 2369 (38)
Statistical Analysis 1: Comparison: Part 1: Normal Renal Function vs Part 1: Mild Renal Impairment; Test type: Other; Ratio of Adjusted Geometric Means = 129.78, 90% CI 2-sided [101.93 to 165.25] — Analysis used one-way ANOVA model with renal function as a fixed effect. The ratio of adjusted geometric means (test [impaired]/reference [normal]) and 90% confidence interval (CI) were expressed as percentages
Statistical Analysis 2: Comparison: Part 1: Normal Renal Function vs Part 1: Moderate Renal Impairment; Test type: Other; Ratio of Adjusted Geometric Means = 138.12, 90% CI 2-sided [113.18 to 168.55] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Part 1: Normal Renal Function vs Part 2: Severe Renal Impairment; Test type: Other; Ratio of Adjusted Geometric Means = 148.02, 90% CI 2-sided [111.40 to 196.68] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero (0) to Extrapolated Infinite Time (AUCinf) of PF-07321332
Description: AUCinf was calculated by AUClast + (Clast/kel). AUClast was the area under the plasma concentration-time profile from time 0 to the time of Clast. Clast was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis and kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Part 1 and Part 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose on Day 1
Population: The PK parameter analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest. Here, "Overall Number of Participants Analyzed" signifies number of participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Number analyzed (Participants) | 10 | 8 | 6 | 7
Nanogram*hour per milliliter | 14460 (20) | 17910 (30) | 27110 (27) | 44040 (33)
Statistical Analysis 1: Comparison: Part 1: Normal Renal Function vs Part 1: Mild Renal Impairment; Test type: Other; Ratio of Adjusted Geometric Means = 123.84, 90% CI 2-sided [99.64 to 153.91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Part 1: Normal Renal Function vs Part 1: Moderate Renal Impairment; Test type: Other; Ratio of Adjusted Geometric Means = 187.40, 90% CI 2-sided [148.52 to 236.46] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Part 1: Normal Renal Function vs Part 2: Severe Renal Impairment; Test type: Other; Ratio of Adjusted Geometric Means = 304.49, 90% CI 2-sided [237.60 to 390.21] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Amount of PF-07321332 Excreted Unchanged in Urine Over 48 Hours (Ae48)
Description: Total amount of unchanged drug excreted in the urine over 48 hours.
Time Frame: Part 1 and Part 2: 0 to 48 hours post dose on Day 1
Population: The PK parameter analysis population included all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligram
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Number analyzed (Participants) | 10 | 8 | 8 | 8
Milligram | 31.20 (45) | 42.65 (23) | 30.83 (56) | 18.46 (50)

4. Primary Outcome: Renal Clearance (CLr) of PF-07321332
Description: Renal clearance was calculated as total amount of unchanged drug excreted in the urine over 48 hours (Ae48) divided by area under the plasma concentration-time profile from time 0 to 48 hours post dose.
Time Frame: Part 1 and Part 2: 0 to 48 hours post dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Number analyzed (Participants) | 10 | 8 | 8 | 8
Liters per hour | 2.180 (50) | 2.395 (33) | 1.154 (71) | 0.4398 (73)

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (SAEs), Treatment Emergent Treatment Related AEs and Treatment Emergent Treatment Related SAEs
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. SAE was any untoward medical occurrence that, at any dose resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect; was a suspected transmission via a Pfizer product of an infectious agent was considered serious; other important medical events. TEAEs were events occurred following start of treatment or increased in severity up to maximum of 35 days after last dose. A treatment-related AE was any untoward medical occurrence attributed to the study drug in a participant who received study drug. Relatedness was judged by investigator.
Time Frame: Part 1 and Part 2: Day -1 up to maximum of 35 days after last dose (maximum of 38 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Number analyzed (Participants) | 10 | 8 | 8 | 8
Participants
  TEAEs | 2 | 1 | 1 | 5
  Treatment Emergent SAEs | 0 | 0 | 0 | 1
  Treatment-related AEs | 0 | 0 | 0 | 2
  Treatment-related SAEs | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: The hematology, clinical chemistry and urinalysis tests were included in the laboratory examination. The criteria for hematology evaluation included hemoglobin less than (<) 0.8*lower limit of normal (LLN), hematocrit <0.8*LLN, erythrocytes <0.8*LLN, erythrocyte mean corpuscular hemoglobin <0.9*LLN and lymphocytes <0.8*LLN. The criteria for clinical chemistry evaluation included neutrophils <0.8*LLN, eosinophils greater than (>) 1.2* upper limit of normal (ULN), monocytes >1.2*ULN, urea nitrogen >1.3*ULN, creatinine >1.3*ULN, urate >1.2*ULN, potassium >1.1*ULN and bicarbonate <0.9*LLN. The criteria for urinalysis evaluation included thyrotropin >1.2*ULN, glucose >1.5*ULN, fibrinogen >1.25*baseline, ketones greater than or equal to (>=) 1, urine protein >=1, nitrite >=1 and leukocyte esterase >=1.
Time Frame: Part 1 and Part 2: Day -1 up to maximum of 35 days after last dose (maximum of 38 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Number analyzed (Participants) | 10 | 8 | 8 | 8
Participants | 5 | 4 | 8 | 8

7. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Supine blood pressure, pulse rate, respiratory rate and oral temperature were evaluated in vital signs examination. Clinical significance was judged by investigator.
Time Frame: Part 1 and Part 2: Day -1 up to maximum of 35 days after last dose (maximum of 38 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Number analyzed (Participants) | 10 | 8 | 8 | 8
Participants | 0 | 0 | 0 | 1

8. Secondary Outcome: Number of Participants With Clinically Significant Findings in Physical Examination
Description: A complete physical examination included, at a minimum, head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, and gastrointestinal, musculoskeletal, and neurological systems. Clinical significance was judged by investigator.
Time Frame: Part 1 and Part 2: Day -1 up to maximum of 35 days after last dose (maximum of 38 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Number analyzed (Participants) | 10 | 8 | 8 | 8
Participants | 0 | 1 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant 12-Lead Electrocardiogram (ECG) Abnormalities
Description: A standard 12-lead ECGs utilizing limb leads (with a 10 second rhythm strip) were collected using an ECG machine that automatically calculates the heart rate and measures PR, QT, and QTc intervals and QRS complex. All scheduled ECGs were performed after the participant had rested quietly for at least 5 minutes in a supine position. Clinical significance was judged by investigator.
Time Frame: Part 1 and Part 2: Day -1 up to maximum of 35 days after last dose (maximum of 38 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Number analyzed (Participants) | 10 | 8 | 8 | 8
Participants | 0 | 0 | 0 | 1

10. Secondary Outcome: Plasma Concentration of PF-07321332 at 12 Hours Post Dose (C12)
Time Frame: Part 1 and Part 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10 and 12 hours post-dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Number analyzed (Participants) | 10 | 8 | 8 | 8
Nanogram per milliliter | 341.9 (35) | 438.0 (30) | 785.6 (33) | 1213 (33)

11. Secondary Outcome: Plasma Concentration of PF-07321332 at 24 Hours Post Dose (C24)
Time Frame: Part 1 and Part 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Number analyzed (Participants) | 10 | 8 | 8 | 8
Nanogram per milliliter | 99.10 (35) | 112.8 (55) | 179.1 (108) | 694.2 (42)

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-07321332
Description: Tmax was observed directly from data as time of first occurrence.
Time Frame: Part 1 and Part 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose on Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Number analyzed (Participants) | 10 | 8 | 8 | 8
Hours | 2.000 [1.00 to 4.00] | 2.000 [1.00 to 3.00] | 2.500 [1.00 to 6.00] | 3.000 [1.00 to 6.05]

13. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero (0) to the Time of the Last Quantifiable Concentration (AUClast) of PF-07321332
Description: Area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration was determined by linear/log trapezoidal method.
Time Frame: Part 1 and Part 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Number analyzed (Participants) | 10 | 8 | 8 | 8
Nanogram*hour per milliliter | 14270 (20) | 17770 (30) | 26660 (21) | 39420 (28)

14. Secondary Outcome: Apparent Clearance (CL/F) of PF-07321332 From Plasma
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the plasma. CL/F was calculated by Dose/AUCinf.
Time Frame: Part 1 and Part 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Number analyzed (Participants) | 10 | 8 | 6 | 7
Liters per hour | 6.913 (20) | 5.581 (30) | 3.689 (27) | 2.270 (33)

15. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-07321332
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed. Vz/F was calculated by dose/(AUCinf*kel). kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Part 1 and Part 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Number analyzed (Participants) | 10 | 8 | 6 | 7
Liters | 74.95 (35) | 51.95 (32) | 50.34 (27) | 42.73 (26)

16. Secondary Outcome: Terminal Elimination Plasma Half-life (t1/2) of PF-07321332
Description: t1/2 was calculated by Loge(2)/kel. kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Part 1 and Part 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 hours post-dose on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
Number analyzed (Participants) | 10 | 8 | 6 | 7
Hours | 7.725 (1.8234) | 6.606 (1.5344) | 9.948 (3.4171) | 13.37 (3.3225)

ADVERSE EVENTS:
Time Frame: Part 1 and Part 2: Day -1 up to maximum of 35 days after last dose (maximum of 38 days)
Description: An AE term may be reported as both a serious and non-serious AE, but are distinct events. An AE may be serious for 1 participant and non-serious for another participant, or a participant may have experienced both a serious and non-serious episode of the same event. Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Arm/Group | Part 1: Normal Renal Function | Part 1: Mild Renal Impairment | Part 1: Moderate Renal Impairment | Part 2: Severe Renal Impairment
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/8 | 1/8
Other Adverse Events (participants affected / at risk) | 2/10 | 1/8 | 1/8 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Normal Renal Function (N=10) | Part 1: Mild Renal Impairment (N=8) | Part 1: Moderate Renal Impairment (N=8) | Part 2: Severe Renal Impairment (N=8)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Normal Renal Function (N=10) | Part 1: Mild Renal Impairment (N=8) | Part 1: Moderate Renal Impairment (N=8) | Part 2: Severe Renal Impairment (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT04909853/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT04909853/SAP_001.pdf